CLINICAL TRIAL: NCT03502902
Title: A Phase I, Double-blind, Placebo-controlled, Single Oral Dose, Safety, Tolerability, and Pharmacokinetic Study, Incorporating an Evaluation of the Effect of Food on the Pharmacokinetics of HEC68498 in Healthy Male and Female Subjects
Brief Title: The Safety, Tolerability and Pharmacokinetic Study of HEC68498 in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCD-DHEC68498-17-001
Record Dates: First submitted 2018-04-10; First posted 2018-04-19 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HEC68498 (Experimental): administered once on first day in each Treatment Period， HEC68498 VS placebo 3:1 ratio
  Interventions: Drug: HEC 68498
- placebo (Placebo Comparator): administered once on first day in each Treatment Period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HEC 68498 — HEC68498 is a potent,highly selective inhibitor of class 1 isozymes of phosphoinositide 3-kinase/mammalian(PI3K) and of the mammalian target of rapamycin (mTOR). It has shown good activity against fibrosis and inflammation in vitro and in vivo, with a lower effective dose and better efficacy than pirfenidone and nintedanib.
  Arms: HEC68498
Drug: Placebo — Placebo
  Arms: placebo

SUMMARY:
A Phase I, Double-blind, Placebo-controlled, Single Oral Dose, Safety, Tolerability, and Pharmacokinetic Study, Incorporating an Evaluation of the Effect of Food on the Pharmacokinetics of HEC68498 in Healthy Male and Female Subjects

DETAILED DESCRIPTION:
Single-dose, sequential-group design incorporating a food-effect evaluation. Each subject will participate in 1 treatment period, except for Group 5, where each subject will participate in 2 treatment periods. In each group, 6 subjects will receive HEC68498 and 2 subjects will receive placebo. Subjects in Group 5 will receive the same dose level of HEC68498 (or placebo) in both treatment periods. All doses will be administered either after an overnight fast of at least 8 hours or, for subjects in the food-effect evaluation, approximately 30 minutes after starting a standard high-fat breakfast. The first 2 subjects in each group will be dosed (1 subject receiving HEC68498 and 1 subject receiving placebo) 48 hours prior to the remainder of the subjects. There will be a minimum of 7 days between dose escalations. The washout period for subjects in Group 5 will be determined following review of available PK data.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, of any race, between 18 and 60 years of age, inclusive, at Screening.
2. Body mass index between 18.0 and 32.0 kg/m2, inclusive, at Screening.
3. In good health, determined by no clinically significant findings from medical history,physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [eg, Gilbert's syndrome] is not acceptable) at Screening or Check-in as assessed by the Investigator (or designee).
4. Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception as detailed in Section 6.6.
5. Where doses exceed 10 mg or where the maximum systemic exposure for any individual subject is predicted to exceed that at the NOAEL of the male rat, male subjects must be sterile. For the purposes of this study, sterile male subjects will include those who have had a vasectomy performed at least 90 days prior to the screening visit and have documentation of azoospermia. Virile male subjects will include all males that do not meet the definition of sterile.
6. Able to comprehend and willing to sign an ICF and to abide by the study restrictions.

Exclusion Criteria:

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
2. Fasting blood glucose >110 mg/dL (confirmed with repeat testing).
3. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).
4. History of stomach or intestinal surgery or resection, including cholecystectomy, that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed).
5. History of alcoholism or drug/chemical abuse within 2 years prior to Check-in.
6. Alcohol consumption of >21 units per week for males and >14 units for females. One unit of alcohol equals 12 oz (360 mL) beer, 1½ oz (45 mL) liquor, or 5 oz (150 mL) wine.
7. Positive urine drug screen (including cotinine) at Screening or Check-in, or positive alcohol breath test at Check-in.
8. Positive hepatitis panel and/or positive human immunodeficiency virus test.
9. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days prior to dosing.
10. Use or intend to use any prescription or nonprescription medications/products, including St. John抯 wort, vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations within 14 days prior to dosing,unless deemed acceptable by the Investigator (or designee).
11. Use of tobacco- or nicotine-containing products within 3 months prior to Check-in.
12. Unwilling or unable to abide by the dietary and exercise restrictions .
13. Receipt of blood products within 2 months prior to Check-in.
14. Donation of blood from 56 days prior to Screening, plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening.
15. Poor peripheral venous access.
16. Have previously completed or withdrawn from this study or any other study investigating HEC68498, and have previously received the investigational product.
17. Subjects who, in the opinion of the Investigator (or designee), should not participate in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Adverse event | up to 4 weeks
  To assess the safety and tolerability of single dose administered

SECONDARY OUTCOMES:
AUC0-∞ | up to one week
  area under the concentration versus time curve (AUC) from time zero to infinity
AUC0-t | up to one week
  AUC from time zero to the time of the last quantifiable concentration time zero to the time of the last quantifiable concentration
Cmax | up to one week
  maximum observed plasma concentration
tmax | up to one week
  time of the maximum observed plasma concentration
t½ | up to one week
  apparent terminal elimination half-life
Vz/F | up to one week
  apparent volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: Irene Mirkin, MD, Principal Investigator — Covance
Locations (1):
- Covance Clinical Research Unit, Inc., Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No